CLINICAL TRIAL: NCT05695053
Title: Low Level Laser Therapy Applied in Orthodontic Tooth Movement
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: CMUH110-REC2-138
Record Dates: First submitted 2023-01-13; First posted 2023-01-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Orthodontic Appliance Complication
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with LLLT (Experimental)
  Interventions: Device: Low Level Laser Therapy
- without LLLT (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Low Level Laser Therapy — Low level laser therapy could provide energy to trigger cell differentiation.
  Arms: with LLLT
Other: Placebo — Placebo
  Arms: without LLLT

SUMMARY:
Currently, orthodontic treatment takes 2-3 years.. If we accelerate tooth movement by low energy laser therapy, we could reduce treatment time. Low Level Laser Therapy(LLLT) applied in Orthodontic Tooth Movement, which stimulates formation of osteoclast-like cells expression in vitro. Osteoclast can be served as an index for tooth movement. Increasing the number of osteoclast will increase bone formation and tooth movement. We plan to find a useful clinical protocol to improve the efficiency of orthodontic tooth movement. Test low energy laser in vitro. Find an effective wavelength and irradiation time to stimulate formation of osteoclast. Develop an useful protocol that clinical orthodontist could follow and reduce orthodontic treatment time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral hygiene
* 18 years old
* Patients who required bilateral canine retraction into the extracted premolar

Exclusion Criteria:

* Serious medical history
* Poor oral hygiene
* Previous orthodontic treatment
* Orthognathic surgery or syndromic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Orthodontic tooth movement | 1-6month
  the distance between canine and premolar

SECONDARY OUTCOMES:
bone density after Orthodontic tooth movement | 1-6month
  bone density change around canine

CONTACTS AND LOCATIONS:
Overall Officials: SHENG-FEN HUANG, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Farivar S, Malekshahabi T, Shiari R. Biological effects of low level laser therapy. J Lasers Med Sci. 2014 Spring;5(2):58-62. PMID 25653800